CLINICAL TRIAL: NCT00436527
Title: MetroGel 1% Hydration Study: A Kinetic Regression Study
Brief Title: Assess the Ability of MetroGel 1% to Deliver Moisture to Facial Skin After a Single Application
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Ronald W. Gottschalk, MD / Medical Director, Galderma Laboratories, L.P.
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: US10041
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2008-04

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Metronidazole gel 1%

INTERVENTIONS:
Drug: Metronidazole gel 1% — Applied once to a test site on the right or left cheek (as determined by a randomization design)
  Other Names: MetroGel® 1%

SUMMARY:
This eight-hour kinetic regression clinical study was conducted to assess the ability of MetroGel® 1% to deliver moisture to facial skin after a single application.

DETAILED DESCRIPTION:
This eight-hour kinetic regression clinical study was conducted to assess the ability of MetroGel® 1% to deliver moisture to facial skin after a single application as measured by the Corneometer CM 825.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe rosacea, defined as the presence of at least moderate erythema with telangiectasia and a minimum of two inflammatory lesions

Exclusion Criteria:

* Individuals with active symptoms of allergy (mild active seasonal allergies are acceptable) or atopic dermatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Six replicate Corneometer CM 825 measurements | 8 hours

SECONDARY OUTCOMES:
Adverse events | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma Laboratories, LP
Locations (1):
- Colorado Springs Research Center, Colorado Springs, Colorado, United States